CLINICAL TRIAL: NCT02451059
Title: Reducing Socioeconomic Disparities in Health at Pediatric Visits
Acronym: WECARE01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Center for Community Health Education Research and Service, Inc. (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-33061; 1R01MD007793-01A1 (NIH)
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Asthma; Obesity; Health Care Utilization; Health Care Disparities; Basic Unmet Social Needs; Blood Pressure; Child Maltreatment; Child Development
Keywords: community resource; well-child care visit; low-income
MeSH Terms: conditions — Asthma; Obesity; Patient Acceptance of Health Care | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-WE CARE (Experimental): 1. The WE CARE survey is used to identify unmet material needs; it will be administered with patient's developmental screening forms at all health supervision visits from birth to two years of age.
  2. Providers will be trained to review the WE CARE survey at health supervision visits and generate our WE CARE community resource handouts (referrals) through the EMR.
  3. A peer patient navigator will offer personalized guidance to families with accessing community resources. The patient navigator will be available for at least a 1/2 day per week at each intervention health center to meet with families and offer guidance. Providers can communicate the patient navigator to refer families via the electronic medical record and families will also have the opportunity to contact the peer navigator at any time via the hotline number listed on the referral information sheets.
  Interventions: Behavioral: WE CARE survey; Behavioral: WE CARE Community Resource Handout; Behavioral: Patient Navigator
- Control-Standard of Care (No Intervention): Participants in the delayed-intervention control group will receive standard pediatric care. However, since the health centers share a common EMR, and for ethical reasons, investigators will also embed the health IT referral mechanism into the EMR at the control sites. Control providers will be made aware of this prior to the start of the study. Although this may potentially reduce the effect size, the investigator's prior study found that the impact on referral rates of provider access to resource information was minimal. Families at control health centers will not receive the WE CARE surveys at health supervision visits and will not have access to the peer patient navigators

INTERVENTIONS:
Behavioral: WE CARE survey — The WE CARE survey, consists of 14 questions used to identify seven unmet material needs (education, employment, food security, housing, childcare, household heat, language). The survey will be administered with patient's developmental screening forms at all health supervision visits from birth to two years of age. The office staff will instruct parents to give the WE CARE survey, along with the developmental screening tool, to their child's provider at the visit.
  Arms: Intervention-WE CARE
Behavioral: WE CARE Community Resource Handout — Providers will be trained to review the WE CARE survey at health supervision visits and generate referrals thru the EMR. Specifically, they will receive a one-hour teaching session one week prior to the study implementation. The goals for the session will include providing an overview of pediatric practice guidelines, introducing the WE CARE survey, reviewing the referral process, and discussing the role of peer patient navigators. Study staff will conduct periodic booster sessions; study staff will also train new providers should there be staff turnover
  Other Names: Resource Referral
  Arms: Intervention-WE CARE
Behavioral: Patient Navigator — The peer patient navigator will offer guidance to families with accessing community resources. They will be available at least .5 days per week at intervention health centers to meet with families and offer guidance as well as be available via a hotline number. The navigator will speak with families and offer guidance on community resources and offer assistance with completing applications. In addition, they will offer to schedule and, if desired, accompany parents to the agencies. Interpreter services will be utilized at the health centers in case the navigator does not speak the parent's language. The navigator will also place an update note in the EMR within 1-month post-visit and one week after any contact with families.
  Arms: Intervention-WE CARE

SUMMARY:
This research project is aimed to assess the effectiveness and impact of a pediatric-based intervention aimed at reducing low-income families' unmet material needs (food, housing, employment, childcare, household heat, education and learning the English language ) on child health.

DETAILED DESCRIPTION:
This project builds upon the PI's prior studies including a recently completed cluster randomized controlled trial (RCT) at community health centers in Boston, which demonstrated a positive impact on provider referrals, discussion, and family receipt of resources.

This study will specifically test the effectiveness of a further strengthened intervention "WE CARE 2.0" on provider referrals and family receipt of resources, along with its impact on child health, health care utilization, and developmental outcomes. Finally, we will gather information from stakeholders at the health centers in order to learn more about the facilitators and barriers to implementation of the model.

The study will take place at six community health centers in the Greater Boston area. The centers will be randomized to either an intervention or control site. Data will be collected on referrals, receipt of resources, and child outcomes from the child's electronic medical record (EMR) from birth to age 3. Focus groups will be used to gather implementation data from intervention health center personnel.

The WE CARE 2.0 intervention consists of: 1) WE CARE surveys which parents complete prior to their child's well-child visits; 2) information technology (IT) generated provider referrals which providers use to provide families with resource information sheets; 3) peer patient navigators who assist families in connecting to available resources and updating providers; and 4) training sessions for providers and office staff.

Families attending the control health centers will receive standard of care. Of note, since the health centers share a common EMR and for ethical reasons, control sites will have access to the IT generated referral mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Child is on Medicaid insurance
* Is attending routine newborn visit

Exclusion Criteria:

* Premature (less than or equal to 32 weeks GA)
* Has a chronic disease
* Has Neonatal Abstinence Syndrome
* Has a foster parent

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1205 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Health care utilization | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will measure whether child is up to date with well child visits between 0-3 years of age. Investigators will measure whether child is up to date on their immunizations between 0-3 years of age. Investigators will measure if and how many times child has been hospitalized or had a visit to the emergency department (ED) between 0-3 years of age.

SECONDARY OUTCOMES:
Child maltreatment | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will measure in the child's EMR whether or not there are any reports of child maltreatment and/or involvement with the Department of Child and Families, at any point, from age 0-3 years of age.
Developmental delay | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will measure whether a developmental delay has been added to the child's problem list in their EMR or if provider has noted a concern of a developmental delay in their routine well-child care notes, at any point, from age 0-3 years of age.
Obesity | Measured at 2-year, 30-month, and 3-year well child care visits (as recommended by the American Academy of Pediatrics)
  Investigators will record the child's reported BMI at their 2-year, 30-month, and 3-year well child care visits from the EMR
Asthma | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will record whether asthma or concerns about asthma have been added to child's problem list in the EMR or noted in the EMR by child's provider at any point, from age 0-3 years of age.
Blood pressure | Measured at 3-year well child care visits
  We will record the child's reported blood pressure number as measured at their 3-year well child care visit. We will gather this information from the EMR.
Provider referrals | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will measure if and how many times a provider made a referral/printed out a community resource handout for patients during their enrollment in the study at any point, from age 0-3 years of age.
Family receipt of community based resource | Throughout child's enrollment in study (0 years through 3 years of age)
  Investigators will determine whether families who were printed out community resource handouts had been able to receive services from a community based resource organization. This will be recorded in the EMR by the patient navigator at anytime from age 0-3 years of age.
Focus group data gathered by audio recordings then transcribed and coded | During 1st month pilot phase and again after investigators have enrolled our the cohort, approximately 3 years after the first focus groups and the study initiation
  Investigators will gain insight into the context and implementation of the augmented WE CARE model from providers and administrative staff at the intervention sites

CONTACTS AND LOCATIONS:
Overall Officials: Arvin Garg, MD MPH, Principal Investigator — Boston University
Locations (6):
- United States (6):
  - South End Community Health Center, Boston, Massachusetts
  - Dorchester House Multi-Service Center, Boston, Massachusetts
  - Codman Square Health Center, Boston, Massachusetts
  - Uphams Corner Health Center, Dorchester, Massachusetts
  - Mattapan Community Health Center, Mattapan, Massachusetts
  - Greater Roslindale Medical and Dental Center, Roslindale, Massachusetts

IPD SHARING:
Plan to Share IPD: No